CLINICAL TRIAL: NCT00285116
Title: The Correlation Between Fasicitis Plantaris and Hallux Rigidus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004/204
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Hallux Rigidus; Fasicitis Plantaris
MeSH Terms: conditions — Hallux Rigidus | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Clinical examination and radiological evaluation

SUMMARY:
Comparison between 3 groups:

* group I has hallux rigidus. Is fasicitis plantaris present?
* group II has fasicitis plantaris. Does the hallux have limited mobility?
* group III does not have hallux rigidus or fasicitis plantaris

ELIGIBILITY:
Inclusion Criteria:

* Hallux rigidus or fasicitis plantaris or healthy volunteer

Exclusion Criteria:

-

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Objective evidence of hallux rigidus being a cause of fasicitis plantaris.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be